CLINICAL TRIAL: NCT03646981
Title: Evaluation of Antibody Detection Tests for Visceral Leishmaniasis Diagnosis in Eastern Africa
Acronym: VL-DX-EAFR
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: University of Gondar (Other); Kenya Medical Research Institute (Other); London School of Hygiene and Tropical Medicine (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: P08002-VL-DX-EAFR
Record Dates: First submitted 2018-08-07; First posted 2018-08-24 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Leishmaniasis, Visceral
Keywords: visceral leishmaniasis; diagnostics; RDT; Eastern Africa
MeSH Terms: conditions — Leishmaniasis, Visceral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Leishmania Ab Rapid Test (CTK, Biotech) — Rapid diagnostic tests to detect antibodies anti-Leishmania
  Other Names: IT Leish (Bio Rad); IgG1 RDT (Coris BioConcept)

SUMMARY:
According to recent estimates by the World Health Organization (WHO) on eastern Africa, not all visceral leishmaniasis (VL) cases reported are confirmed by a laboratory test, probably due to limited access to accurate diagnostic tests and poor reporting. The main approach for VL diagnosis involves antibody detection using the rK39 rapid diagnostic test (RDT) and alternatively the direct agglutination test (DAT) to confirm clinically suspected cases. Suspected cases with negative rK39 RDT and/or DAT results are referred to facilities where examination of tissue aspirate (spleen, bone marrow, lymph node) by microscopy is available. Unfortunately, the diagnostic performance of rK39 in eastern Africa is suboptimal, particularly in settings with a high VL/HIV co-infection rate. A recently developed RDT, based on the recombinant antigen rK28, may overcome this problem, with studies reporting better performance than the rK39. However, data are not definitive, as studies comparing rK28 RDTs with rK39 RDT are limited. Another recently developed RDT detects immunoglobulin G1 (IgG1) specific to Leishmania and has shown promising results in the Indian subcontinent. This study aims to undertake a multi-country assessment of the performance of rK28 and IgG1 RDTs, as compared to the currently used rK39 RDT.

DETAILED DESCRIPTION:
Primary objective and endpoint: To evaluate the performance of different diagnostic tests in detecting anti-Leishmania antibodies to improve early diagnosis of VL in eastern Africa, in particular Ethiopia, and Kenya. Evaluation of the diagnostic performance of the RDTs for primary VL diagnosis based on estimates of sensitivity, specificity, positive and negative predictive values, as well as the degree of agreement between tests.

Design: Prospective single arm diagnostic accuracy study. Multicountry. With participants being suspected cases of VL

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical signs compatible with VL.
* Is a first VL episode suspected.
* Patient ≥ 5 years old (≥ 4 years old in Kenya).
* Patient from whom written informed consent can be obtained or signed by parent or legal guardian if patient is under 18 years of age. In the case of minors, assent from the children (12-17 years old in Ethiopia, Uganda and Sudan, and 13-17 years old in Kenya) will be obtained, as per country legal requirements.
* Clinical samples required VL diagnosis (peripheral blood, lymph node or bone marrow or spleen aspirate) can be obtained from the patient and patient shows willingness.

Exclusion Criteria:

* Patient already on treatment for VL.
* Patient is a suspected VL relapse case.
* Patient has had previous VL episodes.
* Patients < 5 years old (< 4 years old in Kenya).
* Pregnant woman.
* Patient has post/para-kala-azar dermal leishmaniasis (PKDL).

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient reporting to the participating VL treatment centres in Ethiopia, Kenya, Sudan and Uganda and suspected with primary VL is eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 704 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
RDT performance | an average of 1.5 years
  Evaluation of the diagnostic performance of the RDTs for primary VL diagnosis based on estimates of sensitivity, specificity, positive and negative predictive values, as well as the degree of agreement between tests

SECONDARY OUTCOMES:
Time to diagnosis | an average of 1.5 years
  Time taken to perform each diagnostic test, measured from the time the patient reports at the health facility to the time diagnosis is made is established.
New diagnostic algorithm | an average of 1.5 years
  The data generated will be analysed to assess whether the evaluated RDTs can be combined in a new algorithm to improve and accelerate VL diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Israel Cruz, PhD, Principal Investigator — Find
Locations (2):
- Leishmaniasis Research and Treatment Centre, Gondar University Hospital, Gonder, Ethiopia
- Kacheliba District Hospital, Kacheliba, West Pokot County, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing procedures (including data confidentiality) will be carried out in accordance with the regulations defined by IDDO and H2020 Open Research Data Pilot